CLINICAL TRIAL: NCT06072092
Title: Frontal EEG in Out-of-hospital Cardiac Arrest - a Prospective Observational Feasibility Study
Brief Title: Frontal EEG in OHCA Feasibility Study
Acronym: FEICA
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: V2.7.1
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-04

CONDITIONS: Out-Of-Hospital Cardiac Arrest; BIS
Keywords: OHCA; BIS; ROSC; prehospital; PRU
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Out-of-hospital cardiac arrest adult patients: All patients aged ≥18 years and in out-of-hospital cardiac arrest (OHCA) on arrival at the physician response unit (PRU) in Graz, Austria + surroundings.
  Interventions: Device: BIS Monitor

INTERVENTIONS:
Device: BIS Monitor — No interventions will be administered, but in addition to the standard of care according to the Guidelines of the European Resuscitation Council 2021, a frontal EEG-monitoring (BIS), a CPRMeter and a FlowMeter will be installed. The study will be observational only; the readings of the BIS monitor will be blinded to the treating PRU team.

SUMMARY:
This study aims to optimize the treatment of out-of-hospital cardiac arrest (OHCA) by focusing on neurological outcomes through Bispectral Index (BIS) monitoring. It will evaluate the feasibility of BIS monitoring in the prehospital phase, assess the need for sedation based on BIS values, and examine the timing of interventions in ICU (intensive care unit) settings to identify irreversible Hypoxic-Ischemic Brain Injury (HIBI).

DETAILED DESCRIPTION:
The research project is designed to contribute to the low survival discharge rates of OHCA patients in Europe, which is currently around 8%.

Objectives:

1. To assess the feasibility of BIS monitoring in the prehospital environment during CPR and ROSC.
2. To determine the optimal mean BIS cut-off value after ROSC (Return of Spontaneous Circulation) during the prehospital phase.
3. To assess BIS and etCO2 values in OHCA patients under evaluation of CPR quality.
4. To understand the sedation needs based on BIS values.
5. To identify the timing of interventions in the ICU that signify irreversible HIBI.

Phases:

* Phase 1: The initial focus is assessing BIS and etCO2 values in OHCA patients receiving CPR.
* Phase 2: We will investigate whether patients with higher mean BIS values (>25) require earlier and more sedation than those with lower BIS values.
* Phase 3: This phase will examine ICU interventions and their timing to ascertain which patients are at risk of suffering from irreversible HIBI.

Methodology:

The project will utilize prehospital and ICU settings for a multidisciplinary approach, integrating cardiological, neurological, and anesthesiological perspectives. A pilot phase of 5 patients will be conducted initially to fine-tune the protocol and address any technical issues with the equipment.

Timeline:

The study will span approximately 14 months, starting with patient recruitment, data collection, and analysis and ending with the publication of results.

This project aims to provide critical insights into the feasibility and effectiveness of BIS monitoring in improving neurological outcomes for OHCA patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* In out-of-hospital cardiac arrest (OHCA)

Exclusion Criteria:

* BIS application non-possible (for example, due to massive facial trauma)
* No ALS (Advanced Life Support) performed
* Clear signs of death
* Sustained ROSC (>5 minutes after CPR with signs of life) on the arrival of the emergency physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Out-of-hospital cardiac arrest adult patients
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of BIS prehospital via quality parameters. | From PRU arrival until hand-over to the hospital (prehospital phase), on average 60 minutes.
  To evaluate if frontal EEG (BIS) measurements are feasible and valid under CPR and at ROSC in the prehospital setting. The proportion of patients meeting the signal quality criteria in more than 75% of the measurement period (Signal quality index >75, Electromyogram <30) will be presented with a two-sided 95% confidence interval to assess the primary aim.
Feasibility of BIS prehospital via a questionnaire. | Prehospital phase, on average 60 minutes.
  The prehospital BIS feasibility will be assessed with a short questionnaire about the application and its handling.

SECONDARY OUTCOMES:
Prediction of neurological outcome. | Prehospital phase, on average 60 minutes.
  To find the optimal mean BIS cut-off after ROSC throughout the prehospital phase associated with higher CPC scores at 1 month after the event.
CPR quality | Prehospital phase, on average 30 minutes.
  To assess the correlation of BIS and etCO2 values in OHCA patients receiving CPR under evaluation of CPR quality.
Sedation at ROSC | Prehospital phase, on average 30 minutes.
  Patients with higher mean BIS values (>25) will require earlier and more sedation than patients with values below.
ICU care | ICU stay, on average 4 days.
  To assess all timings of interventions on ICU indicating irreversible HIBI.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data will be made available on specific requests.

REFERENCES:
- [Background] Grasner JT, Wnent J, Herlitz J, Perkins GD, Lefering R, Tjelmeland I, Koster RW, Masterson S, Rossell-Ortiz F, Maurer H, Bottiger BW, Moertl M, Mols P, Alihodzic H, Hadzibegovic I, Ioannides M, Truhlar A, Wissenberg M, Salo A, Escutnaire J, Nikolaou N, Nagy E, Jonsson BS, Wright P, Semeraro F, Clarens C, Beesems S, Cebula G, Correia VH, Cimpoesu D, Raffay V, Trenkler S, Markota A, Stromsoe A, Burkart R, Booth S, Bossaert L. Survival after out-of-hospital cardiac arrest in Europe - Results of the EuReCa TWO study. Resuscitation. 2020 Mar 1;148:218-226. doi: 10.1016/j.resuscitation.2019.12.042. Epub 2020 Feb 3. PMID 32027980
- [Background] Sandroni C, Skrifvars MB, Taccone FS. Brain monitoring after cardiac arrest. Curr Opin Crit Care. 2023 Apr 1;29(2):68-74. doi: 10.1097/MCC.0000000000001023. Epub 2023 Feb 16. PMID 36762679
- [Background] Chang CY, Chen CS, Chien YJ, Lin PC, Wu MY. The Effects of Early Bispectral Index to Predict Poor Neurological Function in Cardiac Arrest Patients: A Systematic Review and Meta-Analysis. Diagnostics (Basel). 2020 Apr 30;10(5):271. doi: 10.3390/diagnostics10050271. PMID 32365854
- [Background] Arbas-Redondo E, Rosillo-Rodriguez SO, Merino-Argos C, Marco-Clement I, Rodriguez-Sotelo L, Martinez-Marin LA, Martin-Polo L, Velez-Salas A, Caro-Codon J, Garcia-Arribas D, Armada-Romero E, Lopez-De-Sa E. Bispectral index and suppression ratio after cardiac arrest: are they useful as bedside tools for rational treatment escalation plans? Rev Esp Cardiol (Engl Ed). 2022 Dec;75(12):992-1000. doi: 10.1016/j.rec.2022.03.004. Epub 2022 May 12. English, Spanish. PMID 35570124
- [Derived] Eichinger M, Zoidl P, Reisinger AC, Orlob S, Hatzl S, Eichlseder M, Pichler A, Eberl A, Kuenzer T, Zajic P, Heuschneider L, Honnef G, Rief M, Bornemann-Cimenti H. Assessment of frontal EEG measurement in out-of-hospital cardiac arrest: a prospective observational feasibility study - study protocol. BMJ Open. 2025 Feb 26;15(2):e094258. doi: 10.1136/bmjopen-2024-094258. PMID 40010837